CLINICAL TRIAL: NCT05955638
Title: Management of Myopia in University Students Using Dual Focus Soft Contact Lenses
Acronym: MoMUS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bradford (Other)
Collaborators: University of Huddersfield (Other); CooperVision International Limited (CVIL) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E1060
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Myopia, Progressive
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MiSight dual focus contact lens (Experimental)
  Interventions: Device: MiSight contact lenses
- Proclear single vision contact lens (Active Comparator)
  Interventions: Device: Proclear contact lenses

INTERVENTIONS:
Device: MiSight contact lenses — Contact lens for myopia management.
  Arms: MiSight dual focus contact lens
Device: Proclear contact lenses — Single vision contact lens as control
  Arms: Proclear single vision contact lens

SUMMARY:
The purpose of the study is to quantify the effectiveness of Coopervision MiSight contact lenses in slowing the rate of myopia progression in university students.

DETAILED DESCRIPTION:
MiSight contact lenses have been shown to be a safe and effective way of managing myopia progression in children aged 8-12 years. However, myopic progression is not limited to children of this age group and MiSight lenses have also been shown to be effective in older children aged 11-16 years. There is evidence that progression also occurs in university students. The researchers are therefore investigating the effectiveness of this intervention in a group of UK-based University students.

ELIGIBILITY:
Inclusion Criteria:

* Be a myopic students studying at university
* Be aged 18-21 years at the start of the study
* Show evidence of recent myopia progression prior to commencement of Stage 2 of the study.
* Have read the patient information sheet and be happy to sign the consent forms
* Be willing to adhere to the visit schedule and wearing times described in this protocol
* Agree to lens wearing times of at least 10 hours per day, 6 days per week
* Agree to accept either the control or test lens as assigned by the randomisation
* Have BCVA of +0.10 logMAR or better in each eye

Exclusion Criteria:

* Previous myopia control use (optical or pharmacological)
* Amblyopia
* Ocular pathology such as keratoconus or recurrent corneal infections
* Myopic Rx > 10D
* Astigmatism >1D
* Anisometropia >1.75D
* Binocular Vision anomalies (such as Tropia)
* Medications that affect pupil size or accommodation
* A known allergy to fluorescein or tropicamide
* Biomicroscopic findings that would contraindicate contact lens wear
* The investigator considers that it is not in the best interest of the subject to participate in the study.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in axial length relative to baseline | Baseline, 24 months
Change in spherical equivalent cycloplegic autorefraction relative to baseline | Baseline, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Webber, MOptom, Principal Investigator — University of Bradford; Matthew Cufflin, PhD, Principal Investigator — University of Bradford; Edward Mallen, PhD, Principal Investigator — University of Bradford; Niall Hynes, PhD, Principal Investigator — University of Huddersfield
Locations (2):
- United Kingdom (2):
  - University of Bradford, Bradford, West Yorkshire
  - University of Huddersfield, Huddersfield

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bullimore MA, Brennan NA. Myopia Control: Why Each Diopter Matters. Optom Vis Sci. 2019 Jun;96(6):463-465. doi: 10.1097/OPX.0000000000001367. PMID 31116165
- [Background] Chamberlain P, Peixoto-de-Matos SC, Logan NS, Ngo C, Jones D, Young G. A 3-year Randomized Clinical Trial of MiSight Lenses for Myopia Control. Optom Vis Sci. 2019 Aug;96(8):556-567. doi: 10.1097/OPX.0000000000001410. PMID 31343513
- [Background] Chamberlain P, Bradley A, Arumugam B, Hammond D, McNally J, Logan NS, Jones D, Ngo C, Peixoto-de-Matos SC, Hunt C, Young G. Long-term Effect of Dual-focus Contact Lenses on Myopia Progression in Children: A 6-year Multicenter Clinical Trial. Optom Vis Sci. 2022 Mar 1;99(3):204-212. doi: 10.1097/OPX.0000000000001873. PMID 35086120
- [Background] Jacobsen N, Jensen H, Goldschmidt E. Does the level of physical activity in university students influence development and progression of myopia?--a 2-year prospective cohort study. Invest Ophthalmol Vis Sci. 2008 Apr;49(4):1322-7. doi: 10.1167/iovs.07-1144. PMID 18385044
- [Background] Jorge J, Almeida JB, Parafita MA. Refractive, biometric and topographic changes among Portuguese university science students: a 3-year longitudinal study. Ophthalmic Physiol Opt. 2007 May;27(3):287-94. doi: 10.1111/j.1475-1313.2007.00475.x. PMID 17470242
- [Background] Kinge B, Midelfart A, Jacobsen G, Rystad J. Biometric changes in the eyes of Norwegian university students--a three-year longitudinal study. Acta Ophthalmol Scand. 1999 Dec;77(6):648-52. doi: 10.1034/j.1600-0420.1999.770608.x. PMID 10634556
- [Background] McAlinden C, Pesudovs K, Moore JE. The development of an instrument to measure quality of vision: the Quality of Vision (QoV) questionnaire. Invest Ophthalmol Vis Sci. 2010 Nov;51(11):5537-45. doi: 10.1167/iovs.10-5341. Epub 2010 May 26. PMID 20505205
- [Background] McCullough SJ, O'Donoghue L, Saunders KJ. Six Year Refractive Change among White Children and Young Adults: Evidence for Significant Increase in Myopia among White UK Children. PLoS One. 2016 Jan 19;11(1):e0146332. doi: 10.1371/journal.pone.0146332. eCollection 2016. PMID 26783753
- [Background] Pesudovs K, Garamendi E, Elliott DB. A quality of life comparison of people wearing spectacles or contact lenses or having undergone refractive surgery. J Refract Surg. 2006 Jan-Feb;22(1):19-27. doi: 10.3928/1081-597X-20060101-07. PMID 16447932
- [Background] Ruiz-Pomeda A, Perez-Sanchez B, Valls I, Prieto-Garrido FL, Gutierrez-Ortega R, Villa-Collar C. MiSight Assessment Study Spain (MASS). A 2-year randomized clinical trial. Graefes Arch Clin Exp Ophthalmol. 2018 May;256(5):1011-1021. doi: 10.1007/s00417-018-3906-z. Epub 2018 Feb 3. PMID 29396662
- [Background] Tilia D, Diec J, Ehrmann K, Falk D, Fedtke C, Conrad F, Wu R, Bakaraju RC. Visual Performance and Binocular/Accommodative Function of S.T.O.P. Contact Lenses Compared With MiSight. Eye Contact Lens. 2023 Feb 1;49(2):63-70. doi: 10.1097/ICL.0000000000000950. Epub 2022 Oct 19. PMID 36282205
- [Background] Wolffsohn JS, Kollbaum PS, Berntsen DA, Atchison DA, Benavente A, Bradley A, Buckhurst H, Collins M, Fujikado T, Hiraoka T, Hirota M, Jones D, Logan NS, Lundstrom L, Torii H, Read SA, Naidoo K. IMI - Clinical Myopia Control Trials and Instrumentation Report. Invest Ophthalmol Vis Sci. 2019 Feb 28;60(3):M132-M160. doi: 10.1167/iovs.18-25955. PMID 30817830